CLINICAL TRIAL: NCT04762199
Title: A Phase 1b Safety and Pharmacodynamic Study of MER Tyrosine Kinase Inhibitor, MRX-2843, in Combination With Osimertinib in Advanced EGFR Mutant Non-Small Cell Lung Cancer
Brief Title: MRX-2843 and Osimertinib for the Treatment of Advanced EGFR Mutant Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Conor Steuer, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001681; NCI-2020-08392 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP5153-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH); P50CA217691 (NIH)
Record Dates: First submitted 2021-02-08; First posted 2021-02-21 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — MRX-2843; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (osimertinib, MRX-2843) (Experimental): Patients receive osimertinib PO QD and MRX-2843 PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Flt3/MerTK Inhibitor MRX-2843; Drug: Osimertinib

INTERVENTIONS:
Drug: Flt3/MerTK Inhibitor MRX-2843 — Given PO
  Other Names: MRX 2843; MRX-2843; MRX2843
Drug: Osimertinib — Given PO
  Other Names: AZD-9291; AZD9291; Mereletinib; Tagrisso

SUMMARY:
This phase Ib trial evaluates the best dose and side effects of MRX-2843 when given in combination with osimertinib in treating patients with EGFR gene mutant non-small cell lung cancer that has spread to other places in the body (advanced). MRX-2843 and osimertinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and tolerability of MRX-2843 (MRX-2843) when administered along with osimertinib.

II. Establish the recommended phase 2 dose (RP2D) of the tested combinations.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To perform biomarker profiling in order to identify potential predictive biomarker to optimize treatment efficacy.

OUTLINE: This is a dose-escalation study of MRX-2843.

Patients receive osimertinib orally (PO) once daily (QD) and MRX-2843 PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for minimum of 30 days, or until resolution of treatment-related toxicity to =< grade 1, whichever is longer after removal from study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed metastatic non-small cell lung cancer (NSCLC) with activating EGFR mutation including typical and atypical mutations in egfr exons 19 and 21
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients in the expansion cohort must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Ability to safely swallow oral medication
* Absolute neutrophil count >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 8.5 g/dL (must be > 2 weeks post-red blood cell transfusion)
* Bilirubin =< 1.5 x the upper limit of normal (ULN). For subjects with documented Gilbert's disease, bilirubin =< 3.0 mg/dL. For subjects with documented liver metastases, bilirubin =< 2.5 x ULN
* Serum creatinine =< 1.5 x the ULN or creatinine clearance (CrCl) >= 50 mL/min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x the ULN (=< 5 x the ULN for subjects with liver metastases)
* The effects of MRX-2843 and osimertinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study drug administration
* Females of childbearing potential who are sexually active with a non-sterilized male partner agree to use 2 methods of effective contraception from screening, and agree to continue using such precautions for 90 days after the final dose of study drug; cessation of birth control after this point should be discussed with a responsible physician. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause)
* Non-sterilized males who are sexually active with a female of childbearing potential must agree to use an acceptable method of effective contraception from Day 1 and for 90 days after the final dose of study drug
* Female subjects of childbearing potential must be nonpregnant, and have a negative pregnancy test result at screening and day 1 of cycles 1-6
* Ability to understand and the willingness to sign a written informed consent document
* COHORT SPECIFIC ELIGIBILITY REQUIREMENTS
* Dose Escalation Cohort: Patients with progressive EGFR (+) NSCLC disease; previously treated or naive to EGFR-tyrosine kinase inhibitor (TKI) (previous treatment with 3rd generation EGFR-TKI including osimertinib allowed
* Dose Expansion Cohort A (Treatment naive):

  * Be treatment naive to osimertinib or any other EGFR TKI,
  * If treated with an EGFR TKI in the adjuvant, must have discontinued treatment prior to disease recurrence and be free of recurrence for at least 12 months (+1 day) while off treatment
* Dose Expansion Cohort B (EGFR TKI resistant):

  * Have progression of disease on osimertinib, erlotinib, gefitinib or afatinib as last previous systemic treatment,
  * If not previously treated with osimertinib, must be EGFR-T790M negative as confirmed using a standard testing platform (circulating tumor deoxyribonucleic acid [ctDNA] or tissue based testing) prior to study treatment
* Backfill Cohort C: This cohort will be open to candidates who are not able to get into any of the dose escalation or expansion cohorts. Examples will be a patient already on osimertinib but without disease progression or an otherwise eligible patient who is unable to wait for new cohorts to open due to disease burden and symptoms.

Such patients may be enrolled into the backfill cohort if they meet the following criteria:

* Patients must meet the general eligibility requirements but do not meet cohort specific requirements,
* If currently on osimertinib, must have tolerated the standard dose of 80 mg for at least 2 cycles without any grade > 2 adverse events,
* Will be treated at a dose previously established to be safe from the dose escalation cohort,
* Will not be included in the dose limiting toxicity (DLT) or maximum tolerated dose (MTD) determination,
* Approval by the study sponsor

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1)
* Patients who are receiving any other investigational agents
* Patients with symptomatic untreated brain metastases would be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patient with treated or asymptomatic untreated brain metastasis is allowed on study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MRX-2843 or osimertinib
* Patients with known diagnosis of interstitial lung disease/pneumonitis
* Patients with corrected QT (QTc) interval prolongation > 500 msec (average of 3 readings), family history of congenital long QTc syndrome or torsades
* Patients with known cardiomyopathy or decreased left ventricular ejection fraction (LVEF) < 50%
* Patient with known history of keratitis or symptoms suggestive of keratitis (such as eye inflammation, lacrimation, light sensitivity, blurred vision, eye pain and/or red eye)
* Patients receiving any medications or substances that are inhibitors or inducers of CYP450 enzyme(s) are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because osimertinib is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with osimertinib and MRX-2843, breastfeeding should be discontinued if the mother is treated with the study agents
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with osimertinib and MRX-2843. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Subject has known or suspected history of retinitis pigmentosa or known or suspected familial history of retinitis pigmentosa
* Subject has a history of type 1 diabetes (T1D) or is considered at high risk for T1D, where high risk is defined as

  * Subject has one first-degree relative (defined as parents, offspring or siblings) with T1D and A1C value > 6.5% or subject with two or more first-degree relatives with T1D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2026-12-27 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 3.5 years after study start
  The computation of the dose to be administered to each patient and the 95% highest posterior density credible interval estimate of the MTD will be carried out using computer program escalation with overdose control (EWOC) version 3.1 and R. Upon completion of the trial, the MTD will be estimated as the median of the marginal posterior distribution of the MTD.
Recommended phase 2 dose (RP2D) of the tested combination (dose escalation) | Up to 3.5 years after study start
  The highest dose level of the combination that is under-toxic and safely tolerated would be considered the RP2D.

SECONDARY OUTCOMES:
Predictive Protein Biomarkers | Up to 3.5 years after study start
  Change in the level of expression of biomarkers of interest (phosphorylated and total EGFR)
Predictive Protein Biomarkers | Up to 3.5 years after study start
  Change in the level of expression of biomarkers of interest (phosphorylated and total MERTK)
Overall response rate (ORR) (dose expansion) | Baseline up to the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 3.5 years
  All patients included in the study will be assessed for response to treatment, even if there are major protocol treatment deviations or if they are ineligible.One sample exact binomial test, and logistics regression will be used to test the ORR in the osimertinib resistant cohort.
1-year progression free survival rate (dose expansion) | From start of treatment to time of progression or death, whichever occurs first, assessed at 1 year
  Will be assessed using Kaplan Meier method, log-rank test, and Cox model in the osimertinib naive cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Conor Steuer, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States